CLINICAL TRIAL: NCT03938389
Title: The Role of the Renin-Angiotensin-Aldosterone System in Adiposity, Blood Pressure and Glucose Metabolism Among African Americans: Pilot Study
Brief Title: The Renin-Angiotensin-Aldosterone System in Adiposity, Blood Pressure and Glucose in African Americans
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joshua Joseph, MD, Assistant Professor of Medicine, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2018H0061; K23DK117041 (NIH)
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: PreDiabetes; Impaired Glucose Tolerance; Obesity; Blood Pressure
Keywords: African American; Black; Prediabetes; Impaired Glucose Tolerance
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Obesity | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Intervention Model Description: Randomized prospective controlled clinical trial with three parallel arms, no crossover.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Valsartan (Active Comparator): Valsartan 160 mg twice daily for 26 weeks
  Interventions: Drug: Valsartan 160mg
- Sacubitril/Valsartan (Experimental): Sacubitril/Valsartan (97/103 mg) twice daily for 26 weeks
  Interventions: Drug: Sacubitril-Valsartan Tab 97-103 MG
- Placebo (Placebo Comparator): placebo (+/- amlodipine 2.5-5 mg twice daily if high blood pressure)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sacubitril-Valsartan Tab 97-103 MG — Participants will take Sacubitril-Valsartan for 26 weeks
  Other Names: Entresto
  Arms: Sacubitril/Valsartan
Drug: Valsartan 160mg — Participant will take Valsartan for 26 weeks
  Other Names: Diovan
  Arms: Valsartan
Drug: Placebo Oral Tablet — Participant with take placebo for 26 weeks or if blood pressure elevated will receive standard of care blood pressure medication, amlodipine.
  Arms: Placebo

SUMMARY:
The primary objective is to examine the impact of the Renin-Angiotensin-Aldosterone System (RAAS) blockade with medications (valsartan) or RAAS and neprilysin inhibition (valsartan/sacubitril) vs. placebo on changes in blood sugar and insulin secretion from the pancreas over 26 weeks assessed with glucose clamp studies among African Americans (AAs) with impaired glucose tolerance.

The investigators hypothesize that combined RAAS/neprilysin inhibition will lead to greater improvement in insulin release from the pancreas and improved blood sugar compared to RAAS inhibition alone among AAs with impaired glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* African Americans aged 18-65 years old with a history of impaired fasting glucose, impaired glucose tolerance, hemoglobin A1c 5.7-6.4% or other risk factors for diabetes including metabolic syndrome, family history of type 2 diabetes in the parents or siblings or history of gestational diabetes will be invited to attend a formal screening visit. Participants with impaired glucose tolerance defined as 2-hour plasma glucose 140-199 mg/dl after a fasting 75-g oral glucose tolerance test and who meet other enrollment criteria will be enrolled.

Exclusion Criteria:

* Type 2 Diabetes (American Diabetes Association Criteria)
* Hypertension with systolic blood pressure (SBP) > 150 mmHg or diastolic blood pressure (DBP) > 100 mmHg or taking anti-hypertensive medications
* SBP < 100 mmHg or DBP < 60 mmHg
* Pharmacologic treatment with statins, β-Blockers, angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, renin inhibitors, and/or mineralocorticoid antagonists
* Steroid use
* Hyperkalemia (Potassium > 5.0 milliequivalent/L)
* Abnormal renal function tests: Glomerular Filtration Rate calculated using the Chronic Kidney Disease Epidemiology Equation < 60 ml/min/1.73 m²
* Treatment with oral hypoglycemic medications,
* Use of antipsychotic medications or severe psychiatric disorders (severe mental illness)

Severe Psychiatric Disorders:

* Schizophrenia
* Paranoid and other psychotic disorders
* Bipolar disorders (hypomanic, manic, depressive, and mixed)
* Major depressive disorders (single episode or recurrent)
* Schizoaffective disorders (bipolar or depressive)
* Pervasive developmental disorders
* Obsessive-compulsive disorders
* Depression in childhood and adolescence
* Panic disorder
* Post-traumatic stress disorders (acute, chronic, or with delayed onset)
* Bulimia Nervosa
* Anorexia Nervosa

  * History of, or planned, bariatric surgery,
  * Weight loss > 5% over the previous 6 months,
  * Pregnancy, planning to conceive a child in the next 9 months, or progesterone based contraception and unable to switch to non-progesterone based contraception,
  * Previous or current diagnosis of cardiac structural and functional abnormalities, history or current diagnosis of heart failure (New York Heart Association classes II-IV), history of myocardial infarction, coronary bypass surgery, or percutaneous coronary intervention during the 6 months prior to screening,
  * History of angioedema, or known hypersensitivity to study drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to 26 weeks in β-cell function (first-phase insulin secretion) | 26 weeks
  β-cell function will be assessed by first-phase insulin secretion, calculated as the mean insulin concentration (uIU/mL) over 10 minutes during the hyperglycemic clamp.

SECONDARY OUTCOMES:
Change in Central Aortic Pressure (mmHg) from Baseline to 26 weeks | 26 weeks
  Central Aortic Pressure, measured via a non-invasive method using the SphygmoCor XCEL device, in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Joseph, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No